CLINICAL TRIAL: NCT04907942
Title: Click's Ecological Momentary Assessment (EMA) and Text Message Intervention for Stress Management (FACE STRESS Study)
Brief Title: Ecological Momentary Assessment and Text Message Intervention for Stress Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DL-FACE-101
Record Dates: First submitted 2021-04-02; First posted 2021-06-01 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Stress, Psychological; Loneliness; Covid19; Stress
Keywords: Stress; Anxiety; Ecological Momentary Assessment; Automated Text Message Intervention
MeSH Terms: conditions — Stress, Psychological; COVID-19; Anxiety Disorders | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 week EMA followed by 2weeks of EMA and automated text messages of stress and coping (Active Comparator): 1 weeks of EMA (2 daily surveys per day waking hours to evaluate momentary affects) plus 2 weeks of EMA in combination of automated text messages delivered twice a day, which content follows constructs from The Transactional Model of Stress and Coping (FACE STRESS)
  Interventions: Other: EMA + EMA and FACE Stress
- Control of EMA alone (Other): 3 weeks of EMA, consisting of 2 surveys per day delivered via text message and email during waking hours to prompt participants to complete the survey.
  Interventions: Other: EMA Alone

INTERVENTIONS:
Other: EMA + EMA and FACE Stress — 1 wk of EMA (2 daily surveys per day delivered during waking hours to evaluate momentary affects) plus 2 weeks of EMA and FACE stress
  Other Names: Ecological Momentary Assessments (EMA) & FACE Stress
  Arms: 1 week EMA followed by 2weeks of EMA and automated text messages of stress and coping
Other: EMA Alone — Three weeks of EMA consisting of 2 daily surveys per day delivered during waking hours to evaluate ecological momentary affects.
  Arms: Control of EMA alone

SUMMARY:
Feasibility and acceptability of an Ecological Momentary Assessment (EMA) compared with an EMA plus automated text message intervention for stress management

DETAILED DESCRIPTION:
The purpose of this study is to evaluate feasibility and acceptability of an Ecological Momentary Assessment (EMA) compared with an EMA plus automated text message intervention for stress management in participants with higher-than-average perceived stress conducted in a remote setting.

Study details include:

Study Duration: 7 months Intervention Duration: 3 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 years or older
2. Must reside in an Eastern Standard Time or Central Standard Time zone
3. Able to read and write in English as demonstrated by review and completion of an Informed Consent Form
4. Own an SMS enabled smartphone
5. Scoring >5 on the 4-item Perceived Stress Scale (reflecting higher-than-average perceived stress)

Exclusion Criteria:

1. Reported cognitive impairment and/or psychiatric disorders of the psychotic spectrum
2. Enrolled in another support study
3. Currently receiving psychotherapy through telehealth
4. PHQ-9 score of 20 or greater.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, MDPhD, FAAN, Study Chair — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1:Active Intervention of 1 wk EMA + 2 Wks EMA Plus FACE Stress: 1 wk of Ecological momentary Assessment (EMA), via text message and email followed by 2 additional wks of Ecological momentary Assessment (EMA) in combination with stress management techniques (FACE stress).
- Arm 2: Control Using EMA Alone: Three weeks of Ecological Momentary Assessment (EMA) consisting of 2 daily surveys per day delivered during waking hours to evaluate ecological momentary affects.
Period: Overall Study
Arm/Group | Arm 1:Active Intervention of 1 wk EMA + 2 Wks EMA Plus FACE Stress | Arm 2: Control Using EMA Alone
Started | 39 | 42
Completed | 39 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1) Active Intervention: 1 wk EMA Plus 2 Wks EMA and FACE Stress: 1 wk EMA plus 2 weeks of EMA in combination with constructs from The Transactional Model of Stress and Coping (FACE Stress)
- 2) Control: EMA Alone: Three weeks of EMA consisting of 2 daily surveys per day during waking hours to evaluate momentary affects
- Total: Total of all reporting groups
Arm/Group | 1) Active Intervention: 1 wk EMA Plus 2 Wks EMA and FACE Stress | 2) Control: EMA Alone | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (11.2) | 33.5 (12.5) | 35 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 15 | 16 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 19 | 24 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed EMA and EMA Plus Text Message Intervention or EMA Intervention Alone.
Description: The main outcome of the FACE STRESS study is to evaluate feasibility of an EMA and EMA plus text message intervention (EMA+), assessed by the number of completed individuals after the initial screening, from zero as worst to all subjects (best)
Time Frame: 3 weeks
Population: Feasibility assessed by the number of eligible individuals after the initial screening
Measure: Count of Participants; unit: Participants
Groups:
- 1 Week EMA Followed by 2weeks of EMA and FACE Stress Technique: 1 weeks of EMA (2 daily surveys per day waking hours to evaluate momentary affects) plus 2 weeks of EMA in combination of automated text messages delivered twice a day, which content follows constructs from The Transactional Model of Stress and Coping (FACE stress)
  EMA + EMA and FACE Stress: 1 wk of EMA (2 daily surveys per day delivered during waking hours to evaluate momentary affects) plus 2 weeks of EMA and FACE stress
Arm/Group | 1 Week EMA Followed by 2weeks of EMA and FACE Stress Technique | Control of EMA Alone
Number analyzed (Participants) | 39 | 42
Participants | 39 | 42

ADVERSE EVENTS:
Time Frame: 3 weeks (Intervention period)
Description: pilot study with text messages and no study drugs administration
Groups:
- Active Intervention; 3wks EMA and FACE Stress on Wks 2-3: 1 weeks of EMA (2 daily surveys per day waking hours to evaluate momentary affects) plus 2 weeks of EMA in combination of automated text messages delivered twice a day, which content follows constructs from The Transactional Model of Stress and Coping (FACE stress)
- 3 Wks EMA Alone: Three weeks of EMA consisting of 2 daily surveys per day during waking hours to evaluate momentary affects.
Arm/Group | Active Intervention; 3wks EMA and FACE Stress on Wks 2-3 | 3 Wks EMA Alone
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/42
Other Adverse Events (participants affected / at risk) | 0/39 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT04907942/Prot_SAP_000.pdf